CLINICAL TRIAL: NCT01484730
Title: A Pilot Study to Evaluate Multi-Spectral Imaging (MI) and Laser Speckle Imaging (LSI) and Multiphoton Microscopy (MPM) During Vascular Occlusion
Brief Title: A Pilot Study to Evaluate Multi-Spectral and Laser Speckle Imaging and Multiphoton Microscopy During Vascular Occlusion
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anthony Joseph Durkin, Associate Researcher, BME & Surgery, Director, Laboratory for Functional Imaging Lab, University of California, Irvine
Other Study IDs: 20118370
Record Dates: First submitted 2011-11-29; First posted 2011-12-02 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Abnormal Vascular Flow
MeSH Terms: interventions — Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vascular Occlusion: Multi-Spectral and Laser Speckle Imaging
  Interventions: Device: Multi-Spectral and Laser Speckle Imaging

INTERVENTIONS:
Device: Multi-Spectral and Laser Speckle Imaging — Changes in skin tissue and blood flow.

SUMMARY:
The purpose of this research is to evaluate and validate the performance of non-invasive imaging modalities for assessment of skin. A pressure cuff occlusion will be used to stimulate blood flow dynamic that these instruments are designed to sense. The researcher currently plan to assess only basic feasibility of the imaging instruments.

DETAILED DESCRIPTION:
The primary reason for including pressure cuff occlusion in this protocol is to test the performance of Multi-Spectral Imaging and Laser Speckle Imaging can measure in the full range of vascular conditions ranging from ischemic (under-perfused or unsaturated) to hyperemic (over-perfused and over-saturated).

1. Modulated Imaging a non-contact optical imaging technology can detect the concentration of total hemoglobin, deoxygenated and oxygenated hemoglobin in absolute amounts in units of millimoles / unit volume of tissue measured.
2. Laser Speckle Imaging a non-contact optical imaging technology consists of a coherent light source, camera, and image acquisition system. This image device can measure and compare relative flow in vasculature at varied time points.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult 18 years and older

Exclusion Criteria:

* Younger than 18 years of age
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from University of California Irvine, student and staff member.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-11; Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Skin blood flow | 4 weeks
  The key factor of interest is measuring the changes in the fluorescence signal of the epidermal cells during the arm occlusion, which will provide information about changes in cellular metabolism during cellular oxygen deprivation. Time series of optical sections (two-dimensional x-y images parallel to the skin surface of about 250x250 µm2) at the same depth will be obtained before, during and after the arm occlusion. The images will be based on two-photon excitation of endogenous fluorophores (NADH). To quantify the fluorescence signal, which will provide information about changes of cellular metabolism, we will use the integrated brightness of each image (same rectangular area for all images) as a measure of the signal. The integrated brightness is defined as the sum of pixels weighted over the brightness values (or gray values) of the pixel. A statistical plan is not appropriate at this stage of the pilot study.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Durkin, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Beckman Laser Institute and Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No